CLINICAL TRIAL: NCT00974597
Title: A Randomized, Prospective Comparison of AWBAT™-D and MEPILEX® AG for Treatment of Donor Sites in Burn Surgery
Brief Title: Comparison of AWBAT™-D and MEPILEX® AG for Treatment of Donor Sites in Burn Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Management Decision
Sponsor: Aubrey Inc. (Industry)
Responsible Party: Stephen Moss/President, Aubrey Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #AW-101008DS
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-12

CONDITIONS: Burn Surgery
Keywords: burn; donor site; treatment of burns; Treatment of Donor Sites
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AWBAT™-D and Mepilex® Ag dressings — Comparison of AWBAT™-D and Mepilex® Ag dressings for treatment of donor sites in burn surgery.

SUMMARY:
The purpose of this study is to examine AWBAT™-D compared to Mepilex® Ag for the treatment of donor sites in burn surgery.

ELIGIBILITY:
Inclusion Criteria:

* Burn wounds requiring skin grafting
* Matched donor sites available
* 1-30% TBSA

Exclusion Criteria:

* Severe inhalation injury
* Pregnancy
* Co-morbidity which may compromise healing
* Known allergy to pork or pork products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Compare rate of healing of donor sites | 6 month follow-up

SECONDARY OUTCOMES:
Compare complication rates | 6 month follow-up
Compare patient reported perception of pain | 6 month follow-up
Compare clinical outcome (scarring) | 6 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Doctors Hospital of Augusta, Augusta, Georgia, United States